CLINICAL TRIAL: NCT02173613
Title: Reduction of the Duration of Antibiotic Guided by Procalcitonin in Infections Lungs of Hospitalized Elderly: a Randomized
Brief Title: Reduction the Duration of Antibiotic Therapy in the Elderly (PROPAGE)
Acronym: PROPAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1120
Record Dates: First submitted 2013-06-20; First posted 2014-06-25 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2016-02

CONDITIONS: Lung Infection
Keywords: infection lung elderly patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Procalcitonine (Experimental): every 2 days, they will receive the dose of PCT and decide to stop antibiotic treatment according to the algorithm 2. They will notify the results of clinical evaluations in the electronics and all adverse event report forms.
  Interventions: Other: procalcitonine
- contrôle (No Intervention): Only clinical reassessments will be conducted and documented. Data on antibiotic will be listed and all adverse events. Data on the PCT from D2 to D4, D6, D8 and D15 output or will not be available to the prescriber.

INTERVENTIONS:
Other: procalcitonine — The recommendations will be based on the level of PCT: 4 levels of advice will be given:
  * It is highly recommended to stop antibiotics if PCT <0.1ng/ml, and the recommended stop if 0.1ng/ml <PCT <0.25 ng / ml.
  * It is recommended to continue treatment if 0.25 ng / ml <PCT ng / ml.
  * Finally, if the initial PCT greater than 10 ng / ml, a stop will be advised in case of reduction to less than 10% of baseline level.
  Arms: Procalcitonine

SUMMARY:
The main objective is to evaluate the interest of the repeated measurement of procalcitonin in patients with pulmonary infection to reduce the duration of antibiotic therapy in comparison with a conventional clinical strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years
* Started antibiotics for a chest infection
* Procalcitonin performed J0 antibiotic treatment
* Person affiliated to the social security

Exclusion Criteria:

* Patients with a documented infection with germs after Listeria spp, Legionella pneumophilia, Mycobacterium tuberculosis
* Patients with a documented infection with a virus or parasite (eg hemorrhagic fever, malaria)
* Patients with endovascular infection associated (endocarditis, pacemaker. Intravascular catheter)
* Patients with lung abscess associated upon entry Patients with a chronic infection associated
* Patients with severe immunosuppression (HIV or transplant)
* Palliative patient
* Death within 24 hours of admission to nursing units.
* Presence of antibiotic treatment for chronic infection.
* Patient under guardianship, curatorship or any other administrative or judicial action or deprivation of the right or freedom
* Patients hospitalized without their consent

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Duration of antibiotic therapy | Success of antibiotic therapy within 45 days of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Gaetan Gavazzi, Principal Investigator — University Clinic of Geriatrics Medicine, Division of Medicine multidisciplinary CHU de Grenoble,
Locations (1):
- University Hospital Grenoble, Grenoble, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Background] Polton D, Sermet C. Le vieillissement de la population va-t-il submerger le système de santé ? Bulletin Epidémiologique Hebdomadaire. 2006; 5-6:49-52.
- [Background] Gaymu J. Aspects démographiques du vieillissement; Bulletin Epidémiologique Hebdomadaire. 2006; 5-6:38-9.
- [Background] Fein AM. Pneumonia in the elderly: overview of diagnostic and therapeutic approaches. Clin Infect Dis. 1999 Apr;28(4):726-9. doi: 10.1086/515218. PMID 10825027
- [Background] van der Steen JT, Ooms ME, van der Wal G, Ribbe MW. Withholding or starting antibiotic treatment in patients with dementia and pneumonia: prediction of mortality with physicians' judgment of illness severity and with specific prognostic models. Med Decis Making. 2005 Mar-Apr;25(2):210-21. doi: 10.1177/0272989X05275400. PMID 15800305
- [Background] High KP. Infection as a cause of age-related morbidity and mortality. Ageing Res Rev. 2004 Jan;3(1):1-14. doi: 10.1016/j.arr.2003.08.001. No abstract available. PMID 15163100
- [Background] El Solh AA, Aquilina AT, Gunen H, Ramadan F. Radiographic resolution of community-acquired bacterial pneumonia in the elderly. J Am Geriatr Soc. 2004 Feb;52(2):224-9. doi: 10.1111/j.1532-5415.2004.52059.x. PMID 14728631
- [Background] Torres OH, Munoz J, Ruiz D, Ris J, Gich I, Coma E, Gurgui M, Vazquez G. Outcome predictors of pneumonia in elderly patients: importance of functional assessment. J Am Geriatr Soc. 2004 Oct;52(10):1603-9. doi: 10.1111/j.1532-5415.2004.52492.x. PMID 15450034
- [Background] Bula CJ, Ghilardi G, Wietlisbach V, Petignat C, Francioli P. Infections and functional impairment in nursing home residents: a reciprocal relationship. J Am Geriatr Soc. 2004 May;52(5):700-6. doi: 10.1111/j.1532-5415.2004.52205.x. PMID 15086648
- [Background] Harbarth S. Nosocomial transmission of antibiotic-resistant microorganisms. Curr Opin Infect Dis. 2001 Aug;14(4):437-42. doi: 10.1097/00001432-200108000-00007. PMID 11964862
- [Background] Fischer JE, Harbarth S, Agthe AG, Benn A, Ringer SA, Goldmann DA, Fanconi S. Quantifying uncertainty: physicians' estimates of infection in critically ill neonates and children. Clin Infect Dis. 2004 May 15;38(10):1383-90. doi: 10.1086/420741. Epub 2004 Apr 29. PMID 15156475
- [Background] Christ-Crain M, Stolz D, Bingisser R, Muller C, Miedinger D, Huber PR, Zimmerli W, Harbarth S, Tamm M, Muller B. Procalcitonin guidance of antibiotic therapy in community-acquired pneumonia: a randomized trial. Am J Respir Crit Care Med. 2006 Jul 1;174(1):84-93. doi: 10.1164/rccm.200512-1922OC. Epub 2006 Apr 7. PMID 16603606
- [Background] Yoshikawa TT. Antimicrobial resistance and aging: beginning of the end of the antibiotic era? J Am Geriatr Soc. 2002 Jul;50(7 Suppl):S226-9. doi: 10.1046/j.1532-5415.50.7s.2.x. PMID 12121517
- [Background] Bonomo RA. Multiple antibiotic-resistant bacteria in long-term-care facilities: An emerging problem in the practice of infectious diseases. Clin Infect Dis. 2000 Dec;31(6):1414-22. doi: 10.1086/317489. Epub 2000 Nov 29. PMID 11096012
- [Background] Rooney PJ, O'Leary MC, Loughrey AC, McCalmont M, Smyth B, Donaghy P, Badri M, Woodford N, Karisik E, Livermore DM. Nursing homes as a reservoir of extended-spectrum beta-lactamase (ESBL)-producing ciprofloxacin-resistant Escherichia coli. J Antimicrob Chemother. 2009 Sep;64(3):635-41. doi: 10.1093/jac/dkp220. Epub 2009 Jun 23. PMID 19549667
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Background] Agarwal G, Awasthi S, Kabra SK, Kaul A, Singhi S, Walter SD; ISCAP Study Group. Three day versus five day treatment with amoxicillin for non-severe pneumonia in young children: a multicentre randomised controlled trial. BMJ. 2004 Apr 3;328(7443):791. doi: 10.1136/bmj.38049.490255.DE. Epub 2004 Mar 16. PMID 15070633
- [Background] Singh N, Rogers P, Atwood CW, Wagener MM, Yu VL. Short-course empiric antibiotic therapy for patients with pulmonary infiltrates in the intensive care unit. A proposed solution for indiscriminate antibiotic prescription. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):505-11. doi: 10.1164/ajrccm.162.2.9909095. PMID 10934078
- [Background] Micek ST, Ward S, Fraser VJ, Kollef MH. A randomized controlled trial of an antibiotic discontinuation policy for clinically suspected ventilator-associated pneumonia. Chest. 2004 May;125(5):1791-9. doi: 10.1378/chest.125.5.1791. PMID 15136392
- [Background] el Moussaoui R, de Borgie CA, van den Broek P, Hustinx WN, Bresser P, van den Berk GE, Poley JW, van den Berg B, Krouwels FH, Bonten MJ, Weenink C, Bossuyt PM, Speelman P, Opmeer BC, Prins JM. Effectiveness of discontinuing antibiotic treatment after three days versus eight days in mild to moderate-severe community acquired pneumonia: randomised, double blind study. BMJ. 2006 Jun 10;332(7554):1355. doi: 10.1136/bmj.332.7554.1355. PMID 16763247
- [Background] Gervaix A, Pugin J. [Usefulness of procalcitonin in adults and children]. Rev Med Suisse. 2005 Mar 30;1(13):872-4, 877. French. PMID 15895929
- [Background] Galetto-Lacour A, Zamora SA, Gervaix A. Bedside procalcitonin and C-reactive protein tests in children with fever without localizing signs of infection seen in a referral center. Pediatrics. 2003 Nov;112(5):1054-60. doi: 10.1542/peds.112.5.1054. PMID 14595045
- [Background] Christ-Crain M, Jaccard-Stolz D, Bingisser R, Gencay MM, Huber PR, Tamm M, Muller B. Effect of procalcitonin-guided treatment on antibiotic use and outcome in lower respiratory tract infections: cluster-randomised, single-blinded intervention trial. Lancet. 2004 Feb 21;363(9409):600-7. doi: 10.1016/S0140-6736(04)15591-8. PMID 14987884
- [Background] Gervaix A, Galetto-Lacour A, Gueron T, Vadas L, Zamora S, Suter S, Girardin E. Usefulness of procalcitonin and C-reactive protein rapid tests for the management of children with urinary tract infection. Pediatr Infect Dis J. 2001 May;20(5):507-11. doi: 10.1097/00006454-200105000-00007. PMID 11368108
- [Background] Harbarth S, Holeckova K, Froidevaux C, Pittet D, Ricou B, Grau GE, Vadas L, Pugin J; Geneva Sepsis Network. Diagnostic value of procalcitonin, interleukin-6, and interleukin-8 in critically ill patients admitted with suspected sepsis. Am J Respir Crit Care Med. 2001 Aug 1;164(3):396-402. doi: 10.1164/ajrccm.164.3.2009052. PMID 11500339
- [Background] Gendrel D, Raymond J, Coste J, Moulin F, Lorrot M, Guerin S, Ravilly S, Lefevre H, Royer C, Lacombe C, Palmer P, Bohuon C. Comparison of procalcitonin with C-reactive protein, interleukin 6 and interferon-alpha for differentiation of bacterial vs. viral infections. Pediatr Infect Dis J. 1999 Oct;18(10):875-81. doi: 10.1097/00006454-199910000-00008. PMID 10530583
- [Background] Chirouze C, Schuhmacher H, Rabaud C, Gil H, Khayat N, Estavoyer JM, May T, Hoen B. Low serum procalcitonin level accurately predicts the absence of bacteremia in adult patients with acute fever. Clin Infect Dis. 2002 Jul 15;35(2):156-61. doi: 10.1086/341023. Epub 2002 Jun 17. PMID 12087521
- [Background] Simon L, Gauvin F, Amre DK, Saint-Louis P, Lacroix J. Serum procalcitonin and C-reactive protein levels as markers of bacterial infection: a systematic review and meta-analysis. Clin Infect Dis. 2004 Jul 15;39(2):206-17. doi: 10.1086/421997. Epub 2004 Jul 2. PMID 15307030
- [Background] Christ-Crain M, Muller B. Biomarkers in respiratory tract infections: diagnostic guides to antibiotic prescription, prognostic markers and mediators. Eur Respir J. 2007 Sep;30(3):556-73. doi: 10.1183/09031936.00166106. PMID 17766633
- [Background] Stolz D, Christ-Crain M, Bingisser R, Leuppi J, Miedinger D, Muller C, Huber P, Muller B, Tamm M. Antibiotic treatment of exacerbations of COPD: a randomized, controlled trial comparing procalcitonin-guidance with standard therapy. Chest. 2007 Jan;131(1):9-19. doi: 10.1378/chest.06-1500. PMID 17218551
- [Background] Schuetz P, Christ-Crain M, Wolbers M, Schild U, Thomann R, Falconnier C, Widmer I, Neidert S, Blum CA, Schonenberger R, Henzen C, Bregenzer T, Hoess C, Krause M, Bucher HC, Zimmerli W, Muller B; ProHOSP study group. Procalcitonin guided antibiotic therapy and hospitalization in patients with lower respiratory tract infections: a prospective, multicenter, randomized controlled trial. BMC Health Serv Res. 2007 Jul 5;7:102. doi: 10.1186/1472-6963-7-102. PMID 17615073
- [Background] Briel M, Schuetz P, Mueller B, Young J, Schild U, Nusbaumer C, Periat P, Bucher HC, Christ-Crain M. Procalcitonin-guided antibiotic use vs a standard approach for acute respiratory tract infections in primary care. Arch Intern Med. 2008 Oct 13;168(18):2000-7; discussion 2007-8. doi: 10.1001/archinte.168.18.2000. PMID 18852401
- [Background] Kristoffersen KB, Sogaard OS, Wejse C, Black FT, Greve T, Tarp B, Storgaard M, Sodemann M. Antibiotic treatment interruption of suspected lower respiratory tract infections based on a single procalcitonin measurement at hospital admission--a randomized trial. Clin Microbiol Infect. 2009 May;15(5):481-7. doi: 10.1111/j.1469-0691.2009.02709.x. Epub 2009 Mar 5. PMID 19416298
- [Background] Nobre V, Harbarth S, Graf JD, Rohner P, Pugin J. Use of procalcitonin to shorten antibiotic treatment duration in septic patients: a randomized trial. Am J Respir Crit Care Med. 2008 Mar 1;177(5):498-505. doi: 10.1164/rccm.200708-1238OC. Epub 2007 Dec 20. PMID 18096708
- [Background] Hochreiter M, Kohler T, Schweiger AM, Keck FS, Bein B, von Spiegel T, Schroeder S. Procalcitonin to guide duration of antibiotic therapy in intensive care patients: a randomized prospective controlled trial. Crit Care. 2009;13(3):R83. doi: 10.1186/cc7903. Epub 2009 Jun 3. PMID 19493352
- [Background] Tang H, Huang T, Jing J, Shen H, Cui W. Effect of procalcitonin-guided treatment in patients with infections: a systematic review and meta-analysis. Infection. 2009 Dec;37(6):497-507. doi: 10.1007/s15010-009-9034-2. Epub 2009 Oct 13. PMID 19826761
- [Background] Caterino JM, Scheatzle MD, Forbes ML, D'Antonio JA. Bacteremic elder emergency department patients: procalcitonin and white count. Acad Emerg Med. 2004 Apr;11(4):393-6. doi: 10.1197/j.aem.2003.10.027. PMID 15064215
- [Background] Stucker F, Herrmann F, Graf JD, Michel JP, Krause KH, Gavazzi G. Procalcitonin and infection in elderly patients. J Am Geriatr Soc. 2005 Aug;53(8):1392-5. doi: 10.1111/j.1532-5415.2005.53421.x. PMID 16078967
- [Background] Dwolatzky T, Olshtain-Pops K, Yinnon AM, Raveh D, Rogowski O, Shapira I, Rotstein R, Berliner S, Rudensky B. Procalcitonin in the elderly: normal plasma concentrations and response to bacterial infections. Eur J Clin Microbiol Infect Dis. 2005 Nov;24(11):763-5. doi: 10.1007/s10096-005-0035-5. No abstract available. PMID 16283216
- [Background] Bignardi GE, Dhar R, Heycock R, Bansal S, Majmudar N. Can procalcitonin testing reduce antibiotic prescribing for respiratory infections? Age Ageing. 2006 Nov;35(6):625-6. doi: 10.1093/ageing/afl054. Epub 2006 Jul 5. No abstract available. PMID 16822805
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Guigoz Y, Vellas B, Garry PJ. Assessing the nutritional status of the elderly: The Mini Nutritional Assessment as part of the geriatric evaluation. Nutr Rev. 1996 Jan;54(1 Pt 2):S59-65. doi: 10.1111/j.1753-4887.1996.tb03793.x. No abstract available. PMID 8919685
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Fine MJ, Auble TE, Yealy DM, Hanusa BH, Weissfeld LA, Singer DE, Coley CM, Marrie TJ, Kapoor WN. A prediction rule to identify low-risk patients with community-acquired pneumonia. N Engl J Med. 1997 Jan 23;336(4):243-50. doi: 10.1056/NEJM199701233360402. PMID 8995086
- [Derived] Gavazzi G, Drevet S, Debray M, Bosson JL, Tidadini F, Paccalin M, de Wazieres B, Celarier T, Bonnefoy M, Vitrat V. Procalcitonin to reduce exposure to antibiotics and individualise treatment in hospitalised old patients with pneumonia: a randomised study. BMC Geriatr. 2022 Dec 14;22(1):965. doi: 10.1186/s12877-022-03658-4. PMID 36517740